CLINICAL TRIAL: NCT03977597
Title: Evaluation of Diaphragmatic Function After Bi-pulmonary Transplantation
Acronym: DIATRIB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A02418-47
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-05

CONDITIONS: Lung Transplant, Diaphragmatic Function
Keywords: lung transplant; diaphragm evaluation; ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A current complication after lung transplantation is diaphragmatic dysfunction. These dysfunction result to several factors: duration of mechanical ventilation, chest tube, atelectasis, denutrition, phrenic nerve injury during surgical dissection… Only monocentric and retrospective studies collected diaphragmatic paralysis after lung transplant are published. The incidence of diaphragmatic paralysis in post-operative lung transplantation varies from 3.2% to 16.8%.

The main hypothesis of the study is to defined the incidence of diaphragmatic dysfunction in post-operative lung transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years old)
* Admitted for intensive care that can be spontaneously ventilated after bi- pulmonary transplantation

Exclusion Criteria:

* Minor patient
* Ventilated patients less than 24 hours
* patients in controlled ventilation

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient in immediate postoperative bi-pulmonary transplantation
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-01-03 (Actual); Primary Completion 2021-01-03 (Estimated); Study Completion 2021-01-03 (Estimated)

PRIMARY OUTCOMES:
incidence of diaphragmatic disorders (paralysis, severe and moderate dysfunction) in the post-operative period of bi-pulmonary transplantation | 21 days
  incidence of diaphragmatic disorders (paralysis, severe and moderate dysfunction) in the post-operative period of bi-pulmonary transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson, France